CLINICAL TRIAL: NCT06937866
Title: Maintenance Zanzalintinib With Oral Etoposide Following High-dose Chemotherapy in Patients With Relapsed Metastatic Germ-cell Tumor
Brief Title: Maintenance Zanzalintinib With Etoposide After HDCT in GCT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Principal Investigator, Jennifer King, Assistant Professor of Clinical Medicine, Indiana University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCCC-0894
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Germ Cell Tumor
Keywords: zanzalintinib; maintenance chemotherapy
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 Dose Escalation (Experimental)
  Interventions: Drug: Zanzalintinib; Drug: Etoposide Capsule
- Phase II Dose Expansion (Experimental): Patients will be added at highest zanzalintinib dose tolerated, 40mg or 60mg.
  Interventions: Drug: Zanzalintinib; Drug: Etoposide Capsule

INTERVENTIONS:
Drug: Zanzalintinib — Two zanzalintinib doses of 40mg and 60mg. The initial starting dose of zanzalintinib will be 40mg. The patients will receive zanzalintinib orally daily continuously for 28 day cycles.
Drug: Etoposide Capsule — Oral daily for 21 days of each 28 day cycle.

SUMMARY:
This is an open label, single arm phase I/II trial of maintenance zanzalintinib in combination with oral etoposide in patients with relapsed GCT treated with HDCT and PBSCT with a safety lead-in cohort in patients with relapsed, refractory metastatic GCT.

DETAILED DESCRIPTION:
This prospective, phase I/II trial will initially enroll 9 patients with relapsed, refractory metastatic disease. Two doses of zanzalintinib will be evaluated for toxicity. The patients will receive zanzalintinib orally daily continuously in combination with oral standard of care etoposide daily for 21 days out of 28 day cycles until time of progression or toxicity. The DLT period is 1 cycle of 28 days. We will employ the Bayesian optimal interval (BOIN) design to find the MTD.

ELIGIBILITY:
Inclusion Criteria:

Phase I:

1. Histological or serological evidence of incurable, refractory or relapsed metastatic germ cell tumor, including seminoma, non-seminoma, and women with ovarian GCTs.
2. Must have received initial cisplatin-based combination chemotherapy AND demonstrated progression following at least one salvage regimen for advanced germ-cell neoplasm and now considered incurable with standard therapies, including further chemotherapy or surgery.

   2.1. "Failure" of prior therapy is defined as: 2.1.1.A >25% increase in the products of the perpendicular diameters of measurable tumor masses during prior therapy which are not amenable to surgical resection.

   2.1.2.The presence of new tumors that are not amenable to surgical resection 2.1.3.An increase in AFP or beta-hcg (two separate determinations at least one week apart are required if rising tumor markers are the only evidence of failure).

   NOTE: Patients with clinically growing teratoma (normal declining tumor markers and radiographic or clinical progression) should be considered for surgery.
3. Subjects with relapsed primary mediastinal non-seminomatous germ-cell tumor (PMNSGCT) or late relapse (>2 years) not amenable to resection are eligible if they have received first line platinum-based chemotherapy and are deemed not amenable to surgical resection.

Phase II:

1. Histological or serological evidence of non-seminomatous GCT
2. Relapsed disease after first-line cisplatin-based combination chemotherapy
3. Completed salvage treatment with HDCT and PBSCT for 2 tandem cycles per Institutional Guidelines
4. HDCT must have been used as the initial salvage chemotherapy regimen (2nd line therapy) 4.1. Note: 1 or 2 cycles of standard course regimens prior to HDCT are acceptable (regimens including VeIP [vinblastine+ifosfamide+cisplatin] or TIP [paclitaxel+ifosfamide+cisplatin] or PVB [cisplatin+vinblastine+bleomycin]
5. Normal or declining tumor markers (AFP and hCG) at time of screening per discretion of treating physician. Patients need to be considered disease free with no known active residual GCT.
6. Last dose of HDCT must be ≤ 16 weeks from study registration
7. Women with ovarian germ cell tumors are eligible

For All Patients:

1. Written informed consent and HIPAA authorization for release of personal health information.
2. Capable of understanding and complying with the protocol requirements.
3. Age ≥ 18 years at the time of consent.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 within 28 days of study registration
5. Adverse events from prior therapy recovered to CTCAE v5.0 grade ≤ 2 at time of registration unless AE(s) are clinically nonsignificant and/or stable on supportive therapy (eg, physiological replacement of corticosteroid).
6. Adequate laboratory values obtained within 14 days prior to registration for protocol therapy and as defined below:

   6.1. Hemoglobin ≥ 9g/dL 6.2. WBC ≥ 2500/µL 6.3. Absolute neutrophil count ≥ 1500/mm3 6.4. Platelet count ≥ 100,000/mm3 6.5. Total bilirubin ≤ 1.5 X ULN except patients with documented Gilbert's syndrome (≤ 3 X ULN) 6.6. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤3 X ULN; for patients with hepatic metastases, ALT and AST ≤ 5 X ULN. For subjects with documented bone metastasis ALP ≤ 5 X ULN. 6.7. Serum albumin ≥ 2.8g/dL 6.8. (PT)/INR or partial thromboplastin time (PTT) test ≤ 1.5 x upper limit of normal and activated partial thromboplastin time (aPTT) ≤ 1.2 x upper limit of normal (ULN). 6.9. Calculated creatinine clearance

   ≥ 50 mL/min (≥ 0.67 mL/sec) using the Cockcroft Gault equation. 6.10. Urine protein-to-creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol) creatinine.
7. Sexually active fertile subjects and their partners must agree to use highly effective method of contraception (defined in Appendix II) during the course of the study and for the following durations after the last dose of treatment (whichever is later). An additional contraceptive method, such as a barrier method (eg, condom), is required. In addition, men must agree not to donate sperm and women must agree not to donate eggs (ova, oocyte) for the purpose of reproduction during these same periods.

   1. through 186 days after the last dose of zanzalintinib for women of childbearing potential (WOCBP) or through 96 days after the last dose of zanzalintinib for men,
   2. through 180 days for women of childbearing potential (WOCBP) or through 120 days after the last dose of etoposide for men
8. Female subjects of childbearing potential must not be pregnant at screening. Female subjects are considered to be of childbearing potential, and will need a negative pregnancy test, unless one of the following criteria is met: permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. In addition, females < 55 years-of-age must have a serum follicle stimulating hormone [FSH] level > 40 mIU/mL to confirm menopause).

Note: Documentation may include review of medical records, medical examination, or medical history interview by study site staff.

Exclusion Criteria:

Phase I:

1. Patients who have not received greater than or equal to 1 salvage treatment regimens or have further potentially curative treatment options.

Phase II:

1. Relapsed pure seminoma
2. Rising tumor markers (AFP and hCG) at time of screening per discretion of treating physician
3. Patients who completed 2nd cycle of HDCT (time since last dose of HDCT) > 16 weeks ago

For All Patients:

1. Prior treatment with zanzalintinib
2. Receipt of any type of cytotoxic, small molecule kinase inhibitor, biologic, investigational, or other systemic anticancer therapy (including investigational) within 2 weeks before first dose of study treatment.
3. Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
4. Prior hypersensitivity to etoposide which did not recover with supportive care
5. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment. Note: Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of enrollment. Base of skull lesions without definitive evidence of dural or brain parenchymal involvement are allowed.
6. Concomitant anticoagulation with oral anticoagulants (eg, warfarin, direct thrombin inhibitors) and platelet inhibitors (eg, clopidogrel). Note: Subjects must have discontinued oral anticoagulants within 3 days or 5 half-lives prior to first dose of study treatment, whichever is longer.

   Allowed anticoagulants are the following:
   1. Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
   2. Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen.
7. Prior active malignancy is NOT allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical, breast, or prostate cancer, superficial bladder cancer, Gleason < Grade 7 and ≤ T2N0M0 prostate cancers, or other cancer for which the subject has been disease-free for at least three years or at discretion of treating physician.
8. History of psychiatric illness or social situations that would limit compliance with study requirements.
9. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

   9.1. Unstable or deteriorating cardiovascular disorders: 9.1.1. Congestive heart failure New York Heart Association Class 3 or 4, class 2 or higher, unstable angina pectoris, new onset angina, serious cardiac arrhythmias (eg, ventricular flutter, ventricular fibrillation, Torsades de pointes), unstable or deteriorating cardiovascular disorders.

   9.1.2. Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.

   9.1.3. Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before first dose of study treatment.

   9.2. Pulmonary embolism (PE) or deep vein thrombosis (DVT) or prior clinically significant venous events within 3 months before first dose of study treatment. Note: Subjects with a diagnosis of DVT within 6 months are allowed if asymptomatic and stable at screening and are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen. Note: Subjects who don't require prior anticoagulation therapy may be eligible but must be discussed and approved by the Principal Investigator.

   9.3. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation: 9.3.1. Tumors invading the GI-tract from external viscera 9.3.2. Active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, or acute pancreatitis 9.3.3. Acute obstruction of the bowel, gastric outlet, or pancreatic or biliary duct within 6 months before the first dose unless cause of obstruction is definitively managed and subject is asymptomatic 9.3.4. Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment.

   9.3.5. Known gastric or esophageal varices 9.3.6. Ascites, pleural effusion, or pericardial fluid requiring drainage in the last 4 weeks.
10. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose of study treatment.
11. Symptomatic cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation (asymptomatic or radiated lesions allowed).
12. Lesions invading or encasing any major blood vessels including, but not limited to, inferior vena cava, pulmonary artery, or aorta. Note: Subjects with intravascular tumor extension (eg, tumor thrombus in renal vein or inferior V. cava) may be eligible following Principal Investigator approval.
13. Other clinically significant disorders that would preclude safe study participation.

    13.1. Active infection requiring systemic treatment. Note: Prophylactic antimicrobial treatments (antibiotics, antimycotic, antiviral) are allowed.

    13.2. Known infection with acute or chronic hepatitis B or C, known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness except for subjects meeting all of the following criteria: (1) on stable anti-retroviral therapy; (2) CD4+ T cell count ≥ 200/µL; and (3) an undetectable viral load. Note: HIV testing will be performed at screening if and as required by local regulation. Note: To be eligible, participants taking CYP inhibitors (eg, zidovudine, ritonavir, cobicistat, didanosine) or CYP3 inducers (efavirenz) must change to a different regimen not including these drugs 7 days prior to initiation of study treatment. Anti-retroviral therapies (ART) must have been received for at least 4 weeks prior to the first dose. Note: CD4+ T cell counts, and viral load are monitored per standard of care by the local health care provider.

    13.3. Serious non-healing wound/ulcer/bone fracture. Note: non-healing wounds or ulcers are permitted if due to tumor-associated skin lesions.

    13.4. Malabsorption syndrome 13.5. Pharmacologically uncompensated/symptomatic hypothyroidism. 13.6. Moderate to severe hepatic impairment (Child-Pugh B or C). 13.7. Requirement for hemodialysis or peritoneal dialysis. 13.8. History of solid organ or allogeneic stem cell transplant.
14. Major surgery (as defined in Appendix B; eg GI surgery, removal or biopsy of brain metastasis) within 8 weeks before first dose of study treatment. Prior laparascopic surgeries (ie, nephrectomy) within 4 weeks prior to first dose of study treatment. Minor surgery (eg, simple excision, tooth extraction) within 5 days before first dose of study treatment. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible. Note: Fresh tumor biopsies should be performed at least 5 days before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgical procedures, including biopsies, are not eligible.
15. Corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms per electrocardiogram (ECG) within 14 days of study registration.

    Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility.
16. Pregnant or lactating females.
17. Inability to swallow tablets or ingest a suspension either orally or by a nasogastric (NG) or gastrostomy (PEG) tube.
18. Previously identified allergy or hypersensitivity to components of the study treatment formulations.
19. Prior history of myocarditis.
20. Any complementary medications (eg, herbal supplements or traditional Chinese medicines) to treat the disease under study within 2 weeks before first dose of study treatment.
21. Other conditions, which in the opinion of the Investigator, would compromise the safety of the patient or the patient's ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Rate of hematologic toxicity | 28 days
  Rate of hematologic toxicity including neutropenia, anemia, or thrombocytopenia requiring intervention (transfusions or antibiotics)
Phase 1: Rate of non-hematologic toxicity | 28 days
  Rate of non-hematologic toxicity
Phase II: 12-month Progression Free Survival | 12 months
  12-month PFS based on investigator determination of tumor progression (clinical, radiographic, and/or tumor markers including AFP and hCG)

SECONDARY OUTCOMES:
Phase II: 12-month Overall Survival (OS) | 12 months post time of registration
  12-month OS as determined from time of registration to death from any cause
Phase II: Incidence of Adverse Events | Start of treatment until end of treatment safety assessments (up to 2 years)
  Toxicity measured by the NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0 and need for treatment delay, dose reduction, or early discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer King, MD, Principal Investigator — Indiana University Simon Comprehensive Cancer Center
Locations (1):
- Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana, United States